CLINICAL TRIAL: NCT01000675
Title: Gaining Efficacy Long Term: Hydrosoft, an Emerging, New, Embolic Coil (Gel-the-nec)
Brief Title: Registry for Study of Coils in Intracranial Aneurysms
Acronym: Gel-the-nec
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Abbott (Industry); Albany Medical College (Other); Asan Medical Center (Other); Baylor University (Other); Bronson Methodist Hospital (Unknown); Capital Health, Canada (Other); The Cleveland Clinic (Other); Dalhousie University (Other); Fudan University (Other); Fort Sanders Regional Medical Center (Unknown); JFK Medical Center, Florida (Other); Kobe City Medical Center (Unknown); Methodist Research Institute, Indianapolis (Other); Medical University of South Carolina (Other); Providence Health & Services (Other); Scott and White Hospital & Clinic (Other); Stony Brook University (Other); Thomas Jefferson University (Other); Royal University Hospital Foundation (Other); University of California, Los Angeles (Other); University of Florida (Other); University of Maryland (Other); University of Oklahoma (Other); University of Southern California (Other); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, David F. Kallmes, David F Kallmes, MD, Mayo Clinic, Mayo Clinic
Other Study IDs: 09-002933
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Cerebral Aneurysms
Keywords: aneurysm; coils
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The current proposal describes a post-market, clinical registry of HydroSoft, aimed at gaining robust clinical data in a large set of patients to better define the advantages, and potentially, the disadvantages of the HydroSoft, and to inform future randomized trials.

DETAILED DESCRIPTION:
Aim 1. (Primary Outcome) To test the hypothesis that HydroSoft coils lead to diminished rates of aneurysm recurrence relative to bare platinum coils. In order to test this hypothesis, we will compare recanalization or recurrence rates observed in this prospective registry of HydroSoft coils used as finishing coils to historical series of aneurysms treated with bare platinum coils. This registry is designed to achieve 80% power to detect a minimally clinically relevant difference in rates of recurrence between HydroSoft-treated aneurysms compared with bare platinum coils. Based on recent, prospective, randomized trials assessing both bare platinum coils and hydrogel-bearing coils with 25% and 15% recurrence rates, respectively, we predict a recurrence rate of 18% for HydroSoft treated aneurysms. Typically, a "minimally clinically relevant difference" is on the order of a 30% diminution in a given undesirable outcome. As such, the registry is well powered to detect this minimally clinically relevant difference (18% expected recurrence rate for HydroSoft treated coils versus 25% for the historical control group).

Aim 2. (Secondary Outcome 1) To test the hypothesis that the HydroSoft embolic coil can be placed reliably in intracranial, saccular aneurysms, even late in the embolization procedure. Success of this aim is defined as ease of placement of the HydroSoft device, without need for coil removal and subsequent "finishing" with a bare platinum coil.

Aim 3. (Secondary Outcome 2) To test the hypothesis that use of the HydroSoft embolic coil is associated with risks of thromboembolism similar to that with other coil types, on the order of 3-5% or less.

ELIGIBILITY:
Inclusion Criteria:

1. Patient presenting with a ruptured or un-ruptured cerebral aneurysm appropriate for endovascular treatment as determined by the neurovascular team (neurosurgeon/neurointerventionist)
2. Patient age: patients aged between 21 and 90 years will be eligible.
3. Patient HUNT AND HESS Grade 0-3.
4. Patient has given fully informed consent to endovascular coiling procedure or if patient cannot consent for themselves, appropriate written consent has been sought from their next of kin, or from appropriate power of attorney.
5. Aneurysm 3-15mm in maximum diameter.
6. Patient is willing and able to return for follow up angiography or MRA between 6-18 months.
7. The patient has not been previously entered into this registry
8. The aneurysm has not previously been treated (by coiling or clipping).

Exclusion Criteria:

1. Inability to obtain informed consent.
2. Medical or surgical comorbidity such that the patient's life expectancy is less than 1 year.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All people with cerebral aneurysms between the ages of 21 and 90 that are treated with coils.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
We will compare recanalization or recurrence rates observed in this prospective registry of HydroSoft coils used as finishing coils to historical series of aneurysms treated with bare platinum coils. | 6 - 18 months post coiling

SECONDARY OUTCOMES:
HydroSoft embolic coil can be placed reliably in intracranial, saccular aneurysms, even late in the embolization procedure. | 6 - 18 months post coiling

CONTACTS AND LOCATIONS:
Overall Officials: David F Kallmes, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Brinjikji W, Amar AP, Delgado Almandoz JE, Diaz O, Jabbour P, Hanel R, Hui F, Kelly M, Layton KD, Miller JW, Levy E, Moran C, Suh DC, Woo H, Sellar R, Ho B, Evans A, Kallmes DF. GEL THE NEC: a prospective registry evaluating the safety, ease of use, and efficacy of the HydroSoft coil as a finishing device. J Neurointerv Surg. 2018 Jan;10(1):83-87. doi: 10.1136/neurintsurg-2016-012915. Epub 2017 Jan 30. PMID 28138062
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials